CLINICAL TRIAL: NCT02475213
Title: A Phase 1, Open-Label, Dose Escalation Study of MGA271 in Combination With Pembrolizumab and in Combination With MGA012 in Patients With Melanoma, Squamous Cell Cancer of the Head and Neck, Non-Small Cell Lung Cancer, Urothelial Cancer, and Other Cancers
Brief Title: Safety Study of Enoblituzumab (MGA271) in Combination With Pembrolizumab or MGA012 in Refractory Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGA271-03
Record Dates: First submitted 2015-06-16; First posted 2015-06-18 (Estimated); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Melanoma; Head and Neck Cancer; Non Small Cell Lung Cancer; Urothelial Carcinoma
MeSH Terms: conditions — Melanoma; Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (Experimental): Enoblituzumab 3 mg/kg IV weekly plus pembrolizumab 2 mg/kg IV every 3 weeks
  Interventions: Biological: Enoblituzumab Schedule 1; Biological: Pembrolizumab
- Cohort 2 (Experimental): Enoblituzumab 10 mg/kg IV weekly plus pembrolizumab 2 mg/kg IV every 3 weeks
  Interventions: Biological: Enoblituzumab Schedule 1; Biological: Pembrolizumab
- Cohort 3 (Experimental): Enoblituzumab 15 mg/kg IV weekly plus pembrolizumab 2 mg/kg IV every 3 weeks
  Interventions: Biological: Enoblituzumab Schedule 1; Biological: Pembrolizumab
- Cohort 4 (Experimental): Enoblituzumab 15 mg/kg IV plus retifanlimab 375 mg IV every 3 weeks
  Interventions: Biological: Enoblituzumab Schedule 2; Biological: retifanlimab
- Melanoma Cohort (Experimental): Enoblituzumab 15 mg/kg IV weekly plus pembrolizumab 2 mg/kg IV every 3 weeks
  Interventions: Biological: Enoblituzumab Schedule 1; Biological: Pembrolizumab
- Urothelial Cancer Cohort (Experimental): Enoblituzumab 15 mg/kg IV weekly plus pembrolizumab 2 mg/kg IV every 3 weeks
  Interventions: Biological: Enoblituzumab Schedule 1; Biological: Pembrolizumab
- Non-small Cell Cancer (NSCLC) Cohort (Experimental): Enoblituzumab 15 mg/kg IV weekly plus pembrolizumab 2 mg/kg IV every 3 weeks
  Interventions: Biological: Enoblituzumab Schedule 1; Biological: Pembrolizumab
- Squamous Cell Cancer of Head and Neck (SCCHN) Cohort (Experimental): Enoblituzumab 15 mg/kg IV weekly plus pembrolizumab 2 mg/kg IV every 3 weeks
  Interventions: Biological: Enoblituzumab Schedule 1; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Enoblituzumab Schedule 1 — enoblituzumab is administered by IV infusion once per week for up to 51 doses.
  Other Names: MGA271
  Arms: Cohort 1; Cohort 2; Cohort 3; Melanoma Cohort; Non-small Cell Cancer (NSCLC) Cohort; Squamous Cell Cancer of Head and Neck (SCCHN) Cohort; Urothelial Cancer Cohort
Biological: Pembrolizumab — Pembrolizumab is administered by IV infusion every 3 weeks for up to 17 doses.
  Other Names: Keytruda
  Arms: Cohort 1; Cohort 2; Cohort 3; Melanoma Cohort; Non-small Cell Cancer (NSCLC) Cohort; Squamous Cell Cancer of Head and Neck (SCCHN) Cohort; Urothelial Cancer Cohort
Biological: Enoblituzumab Schedule 2 — Enoblituzumab is administered by IV infusion every 3 weeks for up to 17 doses
  Other Names: MGA271
  Arms: Cohort 4
Biological: retifanlimab — Retifanlimab is administered by IV infusion every 3 weeks for up to 17 doses
  Other Names: INCMGA00012; MGA012
  Arms: Cohort 4

SUMMARY:
The purpose of this study is to evaluate the safety of enoblituzumab (MGA271) in combination with Keytruda (pembrolizumab) when given to patients with B7-H3-expressing melanoma, squamous cell carcinoma of the head and neck (SCCHN), non small cell lung cancer (NSCLC), Urothelial Cancer and other B7-H3 expressing cancers. The study will also evaluate what is the highest dose of enoblituzumab that can be given safely when given with pembrolizumab. Assessments will also be done to see how the drug acts in the body (pharmacokinetics (PK), pharmacodynamics) and to evaluate potential anti-tumor activity of MGA271 in combination with pembrolizumab. Safety and efficacy of enoblituzumab in combination with MGA012 (anti-PD-1 monoclonal antibody; also known as INCMGA00012) will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* To enroll on cohorts 1-4, participants must have a histologically-proven, previously treated, unresectable, locally advanced or metastatic mesothelioma, urothelial cancer, thyroid cancer, pancreatic cancer, ovarian cancer, colon cancer, prostate cancer, soft tissue sarcoma, triple negative breast cancer, renal clear cell cancer, melanoma, squamous cell cancer of the head and neck, or non-small cell lung cancer.
* Participants on the melanoma cohort must have progressed on or after at least one anti-PD-L1 or anti- PD-1 containing therapy.
* Participants on the SCCHN cohort must have progressed on or after platinum-based systemic therapy
* Participants on the NSCLC cohort must have progressed on or after first line systemic therapy
* Participants on the urothelial cancer cohort must have received at least one platinum-containing regimen and have progressed on or after an anti-PD-L1 or anti-PD-1 containing therapy
* Measurable disease per RECIST 1.1 criteria
* Easter Cooperative Oncology Group (ECOG) performance status 0 or 1
* Acceptable laboratory parameters and adequate organ reserve.

Exclusion Criteria:

* Patients with a history of symptomatic central nervous system metastases, unless treated and asymptomatic
* Patients with history of autoimmune disease with certain exceptions such as vitiligo, resolved childhood atopic dermatitis, psoriasis not requiring systemic therapy within the past 2 years, patients with history of Grave's disease that are now euthyroid clinically and by lab testing
* History of allogeneic bone marrow, stem cell, or solid organ transplant
* Treatment with systemic cancer therapy or investigational therapy within 4 weeks of first study drug administration; radiation within 2 weeks; corticosteroids (greater than or equal to 10 mg prednisone or equivalent per day) or other immune suppressive drugs within 2 weeks of first study drug administration
* Trauma or major surgery within 4 weeks of first study drug administration
* History of clinically-significant cardiovascular disease; gastrointestinal perforation; gastrointestinal bleeding, acute pancreatitis or diverticulitis within 4 weeks of first study drug administration
* Active viral, bacterial, or systemic fungal infection requiring parenteral treatment within 7 days of first study drug administration
* Known history of hepatitis B or C infection or known positive test for hepatitis B surface antigen or core antigen, or hepatitis C polymerase chain reaction (PCR)
* Known positive testing for human immunodeficiency virus or history of acquired immune deficiency syndrome
* Known hypersensitivity to recombinant proteins, polysorbate 80, or any excipient contained in the drug or vehicle formulation for MGA271 or pembrolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Ward, MD, Study Director — MacroGenics
Locations (20):
- United States (20):
  - Mayo Clinic - AZ, Scottsdale, Arizona
  - Christiana Care Health Services, Inc., Newark, Delaware
  - Mayo Clinic - FL, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Norton Cancer Institute Research Program, Louisville, Kentucky
  - University of Maryland Greenbaum Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - South Texas Accelerated Research Therapeutics, LLC - Midwest, Grand Rapids, Michigan
  - Mayo Clinic - MN, Rochester, Minnesota
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Gabrail Cancer Institute, Canton, Ohio
  - Hospital of the University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburg, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Greenville Health System, Greenville, South Carolina
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aggarwal C, Prawira A, Antonia S, Rahma O, Tolcher A, Cohen RB, Lou Y, Hauke R, Vogelzang N, P Zandberg D, Kalebasty AR, Atkinson V, Adjei AA, Seetharam M, Birnbaum A, Weickhardt A, Ganju V, Joshua AM, Cavallo R, Peng L, Zhang X, Kaul S, Baughman J, Bonvini E, Moore PA, Goldberg SM, Arnaldez FI, Ferris RL, Lakhani NJ. Dual checkpoint targeting of B7-H3 and PD-1 with enoblituzumab and pembrolizumab in advanced solid tumors: interim results from a multicenter phase I/II trial. J Immunother Cancer. 2022 Apr;10(4):e004424. doi: 10.1136/jitc-2021-004424. PMID 35414591

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: enoblituzumab 3 mg/kg IV weekly for up to 51 doses and pembrolizumab 2 mg/kg IV every 3 weeks for up to 17 doses
- Cohort 2: enoblituzumab 10 mg/kg IV weekly for up to 51 doses and pembrolizumab 2 mg/kg IV every 3 weeks for up to 17 doses
- Cohort 3; Melanoma Cohort; Urothelial Cancer Cohort; NSCLC Cohort; SCCHN Cohort: enoblituzumab 15 mg/kg IV weekly for up to 51 doses and pembrolizumab 2 mg/kg IV every 3 weeks for up to 17 doses
- Cohort 4: enoblituzumab 15 mg/kg IV and retifanlimab 375 mg IV every 3 weeks for up to 17 doses.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Melanoma Cohort | Urothelial Cancer Cohort | NSCLC Cohort | SCCHN Cohort | Cohort 4
Started | 6 | 3 | 3 | 17 | 21 | 40 | 44 | 12
Safety Population (Includes all participants receiving at least 1 dose of enoblituzumab.) | 6 | 3 | 3 | 17 | 21 | 40 | 43 | 12
PK Population (Includes all participants where PK samples could be analyzed.) | 6 | 3 | 3 | 17 | 21 | 39 | 42 | 12
Response Evaluable Population (Includes all participants with pre-dose tumor assessment and at least 1 post-dose tumor assessment.) | 6 | 3 | 3 | 15 | 17 | 34 | 35 | 11
Completed | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 0
Not Completed | 6 | 3 | 3 | 16 | 20 | 37 | 43 | 12
Not completed — Adverse Event | 2 | 0 | 0 | 1 | 1 | 4 | 6 | 2
Not completed — Physician Decision | 1 | 1 | 1 | 0 | 0 | 1 | 4 | 0
Not completed — Progressive Disease | 3 | 2 | 2 | 13 | 15 | 25 | 30 | 10
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Melanoma Expansion; Urothelial Cancer Expansion; NSCLC Expansion; SCCHN Expansion: enoblituzumab 15 mg/kg IV weekly for up to 51 doses and pembrolizumab 2 mg/kg IV every 3 weeks for up to 17 doses
- Cohort 4: enoblituzumab 15 mg/kg IV and retifanlimab 375 mg IV every three weeks for up to 17 doses..
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Melanoma Expansion | Urothelial Cancer Expansion | NSCLC Expansion | SCCHN Expansion | Cohort 4 | Total
Number analyzed (Participants) | 6 | 3 | 3 | 17 | 21 | 40 | 43 | 12 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (7.85) | 41.7 (25.38) | 74.7 (14.64) | 62.9 (14.92) | 67.2 (9.24) | 64.8 (8.20) | 62.7 (9.63) | 62.4 (12.09) | 63.8 (11.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 6 | 6 | 18 | 5 | 6 | 47
  Male | 3 | 1 | 2 | 11 | 15 | 22 | 38 | 6 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 6
  Not Hispanic or Latino | 5 | 3 | 3 | 16 | 21 | 37 | 41 | 10 | 136
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 2 | 6 | 3 | 12
  White | 6 | 3 | 3 | 17 | 19 | 36 | 34 | 8 | 126
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 3 | 14 | 19 | 37 | 36 | 9 | 126
  Australia | 0 | 0 | 0 | 3 | 2 | 2 | 7 | 3 | 17
  Canada | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
ECOG Performance Status [Count of Participants; unit: Participants] — The ECOG Performance Status describes patients level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). Lower scores indicate a more self-sufficient level of functioning.
  Participants
    ECOG 0 | 2 | 1 | 1 | 5 | 5 | 8 | 13 | 4 | 39
    ECOG 1 | 4 | 2 | 2 | 10 | 16 | 32 | 29 | 8 | 103
    Not reported | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 3
Height [Mean (Standard Deviation); unit: Centimeters] | 164.34 (10.12) | 168.5 (6.44) | 170.4 (7.66) | 173.0 (10.41) | 173.4 (9.18) | 169.4 (9.62) | 175.3 (6.31) | 167.0 (15.93) | 171.8 (9.72)
Weight [Mean (Standard Deviation); unit: Kilograms] | 73.2 (8.67) | 63.1 (16.14) | 79.0 (4.55) | 81.5 (24.82) | 82.7 (17.63) | 74.4 (17.15) | 75.6 (13.60) | 91.1 (35.44) | 78.0 (19.43)
B7H3 immunohistochemistry status [Count of Participants; unit: Participants]
  Positive | 4 | 1 | 2 | 16 | 15 | 32 | 37 | 9 | 116
  Negative | 0 | 0 | 0 | 0 | 4 | 3 | 5 | 3 | 15
  Unknown | 2 | 2 | 1 | 1 | 2 | 5 | 1 | 0 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT) After Administration of Enoblituzumab and Pembrolizumab or Retifanlimab
Description: Dose-limiting toxicities are severe side effects related to study treatment that may cause dose interruptions, dose reductions, or withdrawal of treatment.
Time Frame: Study Day 1-42, for Cohorts 1-4.
Population: Participants in Cohorts 1-4 are evaluable for DLT during the first 42 days of treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: enoblituzumab 3 mg/kg IV weekly for up to 51 doses plus pembrolizumab 2 mg/kg every 3 weeks for up to 17 doses
- Cohort 2: enoblituzumab 10 mg/kg IV weekly for up to 51 doses and pembrolizumab 2 mg/kg every 3 weeks for up to 17 doses
- Cohort 3: enoblituzumab 15 mg/kg IV weekly for up to 51 doses pembrolizumab 2 mg/kg every 3 weeks for up to 17 doses
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 6 | 3 | 3 | 12
Participants | 1 | 0 | 0 | 0

2. Secondary Outcome: Mean Maximum Concentration of Enoblituzumab
Description: The highest measured concentration of enoblizuzumab in the bloodstream.
Time Frame: Baseline, 1, 4, 24, and 72 hours after the first dose.
Population: All participants who received at least one dose of study treatment, date and time of dose administration and relative PK sample collection are known and have sufficient concentration data to derive the PK parameter. PK parameters are analyzed by the dose received. Participants in Cohort 3 and the Expansion Cohorts were combined since all participants were dosed at 15 mg/kg.
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- Cohort 2: enoblituzumab 10 mg/kg IV weekly for up to 51 doses plus pembrolizumab 2 mg/kg every 3 weeks for up to 17 doses
- Cohort 3 and Expansion Cohorts: enoblituzumab 15 mg/kg IV weekly for up to 51 doses plus pembrolizumab 2 mg/kg every 3 weeks for up to 17 doses
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Expansion Cohorts | Cohort 4
Number analyzed (Participants) | 6 | 3 | 122 | 12
mcg/mL | 223.5 (62.80) | 860.0 (434.1) | 995.4 (294.4) | 580.2 (133.1)

3. Secondary Outcome: Mean Trough Concentration of Enoblituzumab
Description: Trough concentration is the concentration measured before the a subsequent dose of enoblituzumab.
  MGA271 is characterized by a biphasic concentration-time profile and PPK was used to estimate PK parameters at each dose level
Time Frame: At baseline, and Day 7.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Expansion Cohorts | Cohort 4
Number analyzed (Participants) | 6 | 3 | 122 | 12
mcg/mL | 146.2 (48.1) | 551.0 (323.7) | 607.3 (246.4) | 180.2 (88.0)

4. Secondary Outcome: Mean Area Under the Concentration Time Curve (AUC) From Time 0 to Day 7 of Enoblituzumab
Description: AUC is the total body exposure to enoblituzumab MGA271 is characterized by a biphasic concentration-time profile and PPK was used to estimate PK parameters at each dose level
Time Frame: At baseline, 1, 4, 24, 72 hours, and Day 7.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL*day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Expansion Cohorts | Cohort 4
Number analyzed (Participants) | 6 | 3 | 122 | 12
mcg/mL*day | 1207 (363.3) | 4540 (2445) | 5175 (1820) | 5919 (2009)

5. Secondary Outcome: Mean Clearance of Enoblituzumab
Description: Drug clearance is the amount of drug removed from the bloodstream by the body per unit of time.
Time Frame: At baseline, 1, 4, 24, 72 hours, and Day 7.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters per day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Expansion Cohorts | Cohort 4
Number analyzed (Participants) | 6 | 3 | 122 | 12
liters per day | 0.155 (0.032) | 0.154 (0.076) | 0.235 (0.079) | 0.210 (0.108)

6. Secondary Outcome: Mean Volume of Distribution at Steady State of Enoblituzumab in Combination With Pembrolizumab or Retifanlimab
Description: The volume of distribution is related to how much drug is distributed to body tissues, or remains in the bloodstream
Time Frame: At baseline, 1, 4, 24, and 72 and Day 7.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Expansion Cohorts | Cohort 4
Number analyzed (Participants) | 6 | 3 | 122 | 12
liters | 6.053 (0.986) | 4.340 (0.466) | 5.814 (1.357) | 6.299 (1.009)

7. Secondary Outcome: Mean Terminal Half-life of Enoblituzumab in Combination With Pembrolizumab or Retifanlimab
Description: Terminal half-life is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium MGA271 is characterized by a biphasic concentration-time profile and PPK was used to estimate PK parameters at each dose level
Time Frame: At baseline, 1, 4, 24, and 72 and Day 7.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Expansion Cohorts | Cohort 4
Number analyzed (Participants) | 6 | 3 | 122 | 12
days | 29.22 (4.337) | 23.27 (8.001) | 20.05 (6.975) | 26.63 (11.43)

8. Secondary Outcome: Number of Participants That Develop Enoblituzumab Anti-drug Antibodies (ADA)
Time Frame: Every 3 weeks throughout the study, average duration 13 months.
Population: All participants who received at least one dose of enoblituzumab and have at least one ADA sample sufficient for analysis. ADA samples are analyzed by the dose received. Participants in Cohort 3 and the Expansion Cohorts were combined since all participants were dosed at 15 mg/kg.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 and Expansion Cohorts | Cohort 4
Number analyzed (Participants) | 6 | 3 | 124 | 12
Participants
  Negative at baseline and negative post-baseline | 3 | 3 | 99 | 10
  Negative at baseline and positive at least once post-baseline | 1 | 0 | 1 | 1
  Negative at baseline and not done post-baseline | 0 | 0 | 7 | 0
  Positive at baseline and negative post-baseline | 0 | 0 | 7 | 0
  Positive at baseline and positive at least once post-baseline | 1 | 0 | 2 | 0
  Positive at baseline and not done post-baseline | 0 | 0 | 4 | 0
  Not done at baseline and not done post-baseline | 0 | 0 | 2 | 0
  Not done at baseline and negative post-baseline | 1 | 0 | 2 | 1

9. Secondary Outcome: Number of Participants That Develop Retifanlimab ADA
Time Frame: Every 3 weeks throughout the study, average duration 13 months.
Population: All participants who received at least one dose of retifanlimab and have at least one ADA sample sufficient for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4
Number analyzed (Participants) | 11
Participants
  Negative at baseline and negative post-baseline | 11
  Negative at baseline and positive at least once post-baseline | 0

10. Secondary Outcome: Objective Response Rate
Description: The number of participants with a complete response (CR) or partial response (PR) to enoblituzumab in combination with pembrolizumab or retifanlimab RECIST 1.1 criteria.
Time Frame: Six weeks after the first dose, then every 9 weeks throughout study until discontinuation, average 13 months
Population: Analysis performed using Response Evaluable Population that includes participants with baseline tumor assessment and at least 1 post-baseline tumor assessment.. NSCLC and SCCHN cohorts were subdivided by prior exposure to a PD1 or PDL1 inhibitor for the evaluation of efficacy. .
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Groups:
- NSCLC Cohort: PD1/PDL1 Naïve; NSCLC Cohort: PD1/PDL1 Experienced; SCCHN Cohort: PD1/PDL1 Naïve; SCCHN Cohort: PD1/PDL1 Experienced: enoblituzumab 15 mg/kg IV weekly for up to 51 doses and pembrolizumab 2 mg/kg IV every 3 weeks for up to 17 doses
- Cohort 4: enoblituzumab 15 mg/kg IV and retifanlimab 375 mg IV every three weeks up to 17 doses.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Melanoma Cohort | Urothelial Cancer Cohort | NSCLC Cohort: PD1/PDL1 Naïve | NSCLC Cohort: PD1/PDL1 Experienced | SCCHN Cohort: PD1/PDL1 Naïve | SCCHN Cohort: PD1/PDL1 Experienced | Cohort 4
Number analyzed (Participants) | 6 | 3 | 3 | 15 | 17 | 15 | 19 | 16 | 19 | 12
percentage of participants | 0 [0 to 45.9] | 33.3 [0.8 to 90.6] | 0 [0 to 70.8] | 6.7 [0.2 to 31.9] | 5.9 [0.1 to 28.7] | 33.3 [11.8 to 61.6] | 10.5 [1.3 to 33.1] | 31.3 [11.0 to 58.7] | 0 [0 to 17.6] | 16.7 [2.1 to 48.4]

11. Secondary Outcome: ORR Using Immune-related (ir) RECIST Criteria
Description: The number of participants with a complete response (CR) or partial response (PR) to enoblituzumab in combination with pembrolizumab or retifanlimab using irRECIST 1.1 criteria.
Time Frame: Six weeks after the first dose, then every 9 weeks throughout study until discontinuation, average 13 months
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Melanoma Cohort | Urothelial Cancer Cohort | NSCLC Cohort: PD1/PDL1 Naïve | NSCLC Cohort: PD1/PDL1 Experienced | SCCHN Cohort: PD1/PDL1 Naïve | SCCHN Cohort: PD1/PDL1 Experienced | Cohort 4
Number analyzed (Participants) | 6 | 3 | 3 | 15 | 17 | 15 | 19 | 16 | 19 | 12
percentage of participants | 0 [0 to 45.9] | 33.3 [0.8 to 90.6] | 0 [0 to 70.8] | 6.7 [0.2 to 31.9] | 5.9 [0.1 to 28.7] | 33.3 [11.8 to 61.6] | 5.3 [0.1 to 26.0] | 31.3 [11.0 to 58.7] | 0 [0 to 17.6] | 25.0 [5.5 to 57.2]

12. Secondary Outcome: Best Overall Response (RECIST 1.1)
Description: The participants best response to treatment during their study participation. Responses are categorized as CR, PR, stable disease (SD), progressive disease (PD) or not evaluated (NE)
Time Frame: Evaluated at 6 weeks then every 9 weeks throughout the study until discontinuation, average 13 months.
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Groups:
- NSCLC Cohort: PD1/PDL1 Experienced: enoblituzumab 15 mg/kg IV weekly for up to 51 doses and pembrolizumab 2 mg/kg every 3 weeks for up to 17 doses
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Melanoma Cohort | Urothelial Cancer Cohort | NSCLC Cohort: PD1/PDL1 Naïve | NSCLC Cohort: PD1/PDL1 Experienced | SCCHN Cohort: PD1/PDL1 Naïve | SCCHN Cohort: PD1/PDL1 Experienced | Cohort 4
Number analyzed (Participants) | 6 | 3 | 3 | 15 | 17 | 15 | 19 | 16 | 19 | 12
Participants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  PR | 0 | 1 | 0 | 1 | 1 | 5 | 2 | 4 | 0 | 2
  SD | 4 | 0 | 3 | 5 | 8 | 9 | 9 | 4 | 9 | 7
  PD | 1 | 2 | 0 | 9 | 8 | 1 | 8 | 7 | 10 | 3
  NE | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Best Overall Response (irRECIST 1.1)
Description: as for outcome 12
Time Frame: Evaluated at 6 weeks then every 9 weeks throughout the study until discontinuation, average 13 months.
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Melanoma Cohort | Urothelial Cancer Cohort | NSCLC Cohort: PD1/PDL1 Naïve | NSCLC Cohort: PD1/PDL1 Experienced | SCCHN Cohort: PD1/PDL1 Naïve | SCCHN Cohort: PD1/PDL1 Experienced | Cohort 4
Number analyzed (Participants) | 6 | 3 | 3 | 15 | 17 | 15 | 19 | 16 | 19 | 12
Participants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  PR | 0 | 1 | 0 | 1 | 1 | 5 | 1 | 4 | 0 | 3
  SD | 4 | 0 | 3 | 7 | 8 | 10 | 11 | 5 | 10 | 6
  PD | 1 | 2 | 0 | 7 | 8 | 0 | 7 | 6 | 9 | 3
  NE | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Minimum and Maximum Duration of Response (DoR) Per irRECIST 1.1
Description: The duration of response displays the minimum and maximum range in months from the first documented CR or PR until disease progression or death, whichever is first.
Time Frame: Evaluated at 6 weeks then every 9 weeks throughout the study until discontinuation, average13 months.
Population: as for outcome 10
Measure: Number; unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Melanoma Cohort | Urothelial Cancer Cohort | NSCLC Cohort: PD1/PDL1 Naïve | NSCLC Cohort: PD1/PDL1 Experienced | SCCHN Cohort: PD1/PDL1 Naïve | SCCHN Cohort: PD1/PDL1 Experienced | Cohort 4
Number analyzed (Participants) | 6 | 3 | 3 | 15 | 17 | 15 | 19 | 16 | 19 | 12
months
  Minimum DoR | NA — There were no responses in this group. | 25.95 | NA — There were no responses in this group. | 6.14 | 28.89 | 3.48 | 4.44 | 4.17 | NA — There were no responses in this group | 3.45
  Maximum DoR | NA — There were no responses in this group. | 25.95 | NA — There were no responses in this group. | 6.14 | 25.89 | 32.00 | 4.44 | 23.72 | NA — There were no responses in this group | 6.24

15. Secondary Outcome: Minimum and Maximum DoR Per RECIST 1.1
Description: as for outcome 14
Time Frame: Evaluated at 6 weeks then every 9 weeks throughout the study until discontinuation, average 13 months.
Population: as for outcome 10
Measure: Number; unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Melanoma Cohort | Urothelial Cancer Cohort | NSCLC Cohort: PD1/PDL1 Naïve | NSCLC Cohort: PD1/PDL1 Experienced | SCCHN Cohort: PD1/PDL1 Naïve | SCCHN Cohort: PD1/PDL1 Experienced | Cohort 4
Number analyzed (Participants) | 6 | 3 | 3 | 15 | 17 | 15 | 19 | 16 | 19 | 12
months
  Minimum DoR | NA — There were no responses in this group | 25.95 | NA — There were no responses in this group | 6.14 | 25.89 | 3.48 | 4.44 | 4.17 | NA — There were no responses in this group | 3.45
  Maximum DoR | NA — There were no responses in this group | 25.95 | NA — There were no responses in this group | 6.14 | 25.89 | 32.00 | 4.44 | 23.72 | NA — There were no responses in this group | 6.24

16. Secondary Outcome: Median Progression-free Survival (PFS) Using RECIST 1.1
Description: The time from the first infusion of pembrolizumab or retifanlimab until documented disease progression or death from any cause.
Time Frame: Evaluated at 6 weeks then every 9 weeks throughout the study until discontinuation, average 13 months.
Population: PFS was calculated using the safety population. NSCLC and SCCHN cohorts were subdivided by prior exposure to a PD1 or PDL1 inhibitor for the evaluation of efficacy only. Safety assessment was conducted regardless of prior exposure to a PD1 or PDL1 inhibitor.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Melanoma Cohort: enoblituzumab 15 mg/kg IV weekly for up to 51 doses and pembrolizumab 2 mg/kg every 3 weeks for up to 17 doses
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Melanoma Cohort | Urothelial Cancer Cohort | NSCLC Cohort: PD1/PDL1 Naïve | NSCLC Cohort: PD1/PDL1 Experienced | SCCHN Cohort: PD1/PDL1 Naïve | SCCHN Cohort: PD1/PDL1 Experienced | Cohort 4
Number analyzed (Participants) | 6 | 3 | 3 | 17 | 21 | 17 | 23 | 19 | 24 | 12
months | NA [1.41 to NA] — The upper limit of the confidence level was not reached. | 1.4 [1.22 to NA] — The upper limit of the confidence level was not reached. | 3.6 [3.32 to 3.91] | 2.0 [1.38 to 4.83] | 2.2 [1.28 to 5.52] | 5.1 [3.19 to NA] — The upper limit of the confidence level was not reached. | 3.5 [1.41 to 5.75] | 3.5 [1.28 to 13.83] | 1.4 [1.35 to 3.55] | 4.8 [1.38 to 11.96]

17. Secondary Outcome: Median PFS Using irRECIST 1.1 Criteria
Description: as for outcome 16
Time Frame: Evaluated at 6 weeks then every 9 weeks throughout the study until discontinuation, average 13 months.
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Melanoma Cohort | Urothelial Cancer Cohort | NSCLC Cohort: PD1/PDL1 Naïve | NSCLC Cohort: PD1/PDL1 Experienced | SCCHN Cohort: PD1/PDL1 Naïve | SCCHN Cohort: PD1/PDL1 Experienced | Cohort 4
Number analyzed (Participants) | 6 | 3 | 3 | 17 | 21 | 17 | 23 | 19 | 24 | 12
months | NA [1.41 to NA] — The upper limit of the confidence level was not reached. | 1.4 [1.22 to NA] — The upper limit of the confidence level was not reached. | 3.6 [3.32 to 3.91] | 2.0 [1.38 to 4.83] | 2.2 [1.28 to 5.52] | 5.1 [3.19 to NA] — The upper limit of the confidence level was not reached. | 3.5 [1.45 to 5.75] | 3.5 [1.28 to 13.83] | 1.4 [1.35 to 3.55] | 4.8 [1.38 to 11.96]

18. Secondary Outcome: Median Overall Survival
Description: The time from the first infusion of pembrolizumab or retifanlimab until death from any cause.
Time Frame: Evaluated at 6 weeks then every 9 weeks throughout the study until discontinuation, average 13 months.
Population: OS was calculated using the safety population. NSCLC and SCCHN cohorts were subdivided by prior exposure to a PD1 or PDL1 inhibitor for the evaluation of efficacy only. Safety assessment was conducted regardless of prior exposure to a PD1 or PDL1 inhibitor.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Melanoma Cohort | Urothelial Cancer Cohort | NSCLC Cohort: PD1/PDL1 Naïve | NSCLC Cohort: PD1/PDL1 Experienced | SCCHN Cohort: PD1/PDL1 Naïve | SCCHN Cohort: PD1/PDL1 Experienced | Cohort 4
Number analyzed (Participants) | 6 | 3 | 3 | 17 | 21 | 17 | 23 | 19 | 24 | 12
months | 18.0 [7.10 to NA] — The upper limit of the confidence interval was not reached. | 10.3 [7.75 to NA] — The upper limit of the confidence interval was not reached. | 6.3 [5.82 to 6.70] | 14.4 [9.00 to NA] — The upper limit of the confidence interval was not reached. | 5.7 [3.09 to 11.10] | 10.3 [6.28 to 18.50] | 6.0 [2.96 to 10.78] | 17.9 [5.13 to NA] — The upper limit of the confidence interval was not reached. | 6.9 [4.75 to 9.69] | NA [NA to NA] — There were no death events in this cohort by the end of the study. OS and confidence interval could not be calculated.

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of first dose through 28 days after the last dose or until the start of another anti-cancer treatment, average 12 months. All cause mortality was assessed from the time of first dose until death, up to 18 months.
Description: Adverse event are based on physical findings, patient reports, and significant laboratory values.
  Progression of neoplasm causing hospitalization or death is an antitumor activity outcome and not an SAE, unless considered drug-related by the investigator.
  On participant was enrolled in the study and never treated so the safety population and all-cause mortality is 145.
Groups:
- Cohort 4: enoblituzumab 15 mg/kg IV and pembrolizumab 2 mg/kg IV every 3 weeks for up to 17 doses.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Melanoma Cohort | Urothelial Cancer Cohort | NSCLC Cohort | SCCHN Cohort | Cohort 4
All-Cause Mortality (participants affected / at risk) | 4/6 | 2/3 | 2/3 | 11/17 | 16/21 | 33/40 | 30/43 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/3 | 2/3 | 8/17 | 4/21 | 14/40 | 18/43 | 3/12
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 3/3 | 17/17 | 21/21 | 40/40 | 42/43 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=3) | Cohort 3 (N=3) | Melanoma Cohort (N=17) | Urothelial Cancer Cohort (N=21) | NSCLC Cohort (N=40) | SCCHN Cohort (N=43) | Cohort 4 (N=12)
Granulomatous lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis syndrome (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 2 | 6 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral artery thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=3) | Cohort 3 (N=3) | Melanoma Cohort (N=17) | Urothelial Cancer Cohort (N=21) | NSCLC Cohort (N=40) | SCCHN Cohort (N=43) | Cohort 4 (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 4 | 3 | 3 | 7 | 3
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 2 | 4 | 6 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 4 | 13 | 9 | 4
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 7 | 2 | 4 | 8 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 3 | 9 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 4 | 5 | 4 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 4 | 5 | 4 | 0
Fatigue (General disorders) | 2 | 1 | 2 | 7 | 4 | 15 | 19 | 2
Pyrexia (General disorders) | 0 | 1 | 0 | 4 | 4 | 2 | 11 | 2
Chills (General disorders) | 1 | 0 | 0 | 1 | 2 | 3 | 5 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 3 | 2 | 2 | 3 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 6 | 0 | 3 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 9 | 10 | 24 | 16 | 6
Lipase increased (Investigations) | 0 | 0 | 0 | 2 | 2 | 6 | 2 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 7 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 5 | 11 | 5 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 5 | 4 | 0 | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3 | 2 | 5 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 7 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3 | 3 | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 4 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 1 | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 3 | 8 | 4 | 8 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2 | 6 | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 4 | 3 | 3 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 3 | 2 | 3 | 6 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 6 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 1 | 1 | 5 | 3 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 3 | 3 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1 | 4 | 8 | 7 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 2 | 10 | 5 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 5 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 2 | 5 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4 | 1 | 2 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 2 | 3 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 2 | 4 | 5 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT02475213/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT02475213/SAP_001.pdf